CLINICAL TRIAL: NCT01492036
Title: Long-Term Follow-Up Study of Recipients of Gene Transfer Research Protocols
Brief Title: Long-Term Follow-Up of Recipient of Gene Transfer Research
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Cancer Institute (NCI) (NIH); Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2006-0676; R01CA124782 (NIH); R01CA141303 (NIH); NCI-2021-14027 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Retroviridae Infections; Cancer
Keywords: Replication-Competent Retrovirus; RCR; Gene transfer therapy; Registry; Medical information database; Vector or vector-treated cells; Blood draw; Computed tomography; CT; Questionnaires; Surveys; Gene Transfer Research; National Gene Vector Biorepository and Coordinating Center; NGVB
MeSH Terms: conditions — Retroviridae Infections; Neoplasms | interventions — Hematologic Tests; Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Study visits once a year during Years 1-5. Blood (about 2-4 tablespoons each time) drawn for routine tests. If retroviral gene transfer therapy received, blood (up to 4 tablespoons each time) drawn every 3 months for first year after gene transfer therapy and once a year after that. If joining study more than a year after gene transfer therapy, RCR test performed once a year for all 15 years of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gene Transfer Therapy: Study participants receiving gene therapy product at MD Anderson Cancer Center
  Interventions: Other: Blood Tests; Behavioral: Questionnaires

INTERVENTIONS:
Other: Blood Tests — If participant received retroviral gene therapy, blood test performed to check for a type of infection called the replication-competent retrovirus (RCR). Blood (up to 4 tablespoons each time) drawn every 3 months for first year after gene transfer therapy and once a year after that.
  Other Names: Blood draw
Behavioral: Questionnaires — Once a year during Years 1-5, questionnaire completions that asks about medical history (general health, the status of any medical conditions, and any illnesses or hospitalizations that may have occurred). It should take about 15-30 minutes to complete.
  Once a year during Years 6-15, completion of mailed questionnaire. Participant will be asked about medical history (including if participant has had any children since the infusion) and whether there have been any changes in contact information. The questionnaires should take about 15-30 minutes each time.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to collect information about the long-term safety of gene transfer therapy. This study is also designed to create a database of medical information about patients who have received gene transfer therapy, in order for researchers to track and review the long-term safety and any effects (good or bad) of gene transfer therapy.

DETAILED DESCRIPTION:
Study Procedures for Years 1-5:

If you agree to take part in this study, you will come to the clinic for study visits once a year during Years 1-5. It is your choice whether to visit your regular local doctor or your study doctor at MD Anderson. (If you visit your regular local doctor, you will need to have your test results and blood samples mailed to the study staff.) You will receive a reminder phone call once a year, when it is time to schedule these visits.

At these visits, the following procedures will be performed:

* Blood (about 2-4 tablespoons each time) will be drawn for routine tests.
* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate).
* You will fill out a questionnaire that asks about your medical history (your general health, the status of any medical conditions, and any illnesses or hospitalizations that may have occurred). It should take about 15-30 minutes to complete.
* You will be asked if there have been any changes in your contact information.
* If necessary to check the status of the disease, you will have scans (x-rays and/or computed tomography [CT] scans) and/or additional routine blood tests (about 1-2 tablespoons).

Study Procedures for Years 6-15:

Once a year during Years 6-15, the research staff will contact you. Either over the phone, by email, or by mail (but usually by mail, with an enclosed questionnaire), you will be asked about your medical history (including if you have had any children since the infusion) and whether there have been any changes in your contact information. The phone calls and questionnaires should take about 15-30 minutes each time.

Results of Study Testing:

If any of the tests that are performed in this study suggest that you may have a medical condition and/or side effect that is likely to be related to the gene transfer therapy, the study doctor will contact you. You will receive a referral in case you would like to seek medical care for the condition and/or side effect.

You and/or your insurance provider will be responsible for the costs of any CT scans and x-rays that may be needed for this study.

Study Database:

Your medical information that is collected for this study will be stored in a research database at MD Anderson for use in future research related to the safety and effects of gene transfer therapy.

Your data will be given a code number. No identifying information will be directly linked to your data. Only the researcher or authorized personnel in charge of the database will have access to the code numbers and be able to link the data to you. This is to allow medical information related to your data to be updated as needed. Other researchers using your data will not be able to link this data to you.

Changes in Parent/Guardian Contact:

If you are younger than 18 years old when joining this study but turn 18 during this study, starting then, the research staff will contact you directly for this study instead of your parent/guardian. However, if you would prefer for your parent/guardian to still be the main contact person, please tell the study staff.

Length of Study Participation:

After 15 years, your participation in this study will be over unless the FDA decides that follow-up must continue.

This is an investigational study.

Up to 130 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or patient's legal representative(s) provided written informed consent to participate in a gene transfer study at the University of Texas MD Anderson Cancer Center (MD Anderson).
2. Patient will receive vector or vector-treated cells at MD Anderson.
3. Patient or patient's legal representative(s) is/are able to provide written informed consent to participate in this long-term follow-up protocol for gene transfer participants for up to 15 years following administration of gene therapy product.
4. Agree to allow clinical samples to be collected and stored at MD Anderson and/or at a NIH designated facility such as the NGVB.

Exclusion Criteria:

1) Subject's gene transfer protocol is not approved at MD Anderson Cancer Center.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Gene transfer therapy in an M. D. Anderson Cancer Center research study in Houston, Texas
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2011-12-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Document Long-Term Safety of Gene-Transfer Research | 15 years
  First 5 years following infusion of vector or vector-treated cells: Participants evaluated on annual basis. Years 6 to 15 following infusion of vector or vector-treated cells: Participants mailed questionnaires. Participants in retroviral studies: Up to 60 mL (max 1 mL/kg) blood will be obtained to check for replication-competent retrovirus (RCR) every 3 months during the first year, and then blood archived annually thereafter. Replication competent vector testing performed when there is a clinical indication or when requested by the FDA.

CONTACTS AND LOCATIONS:
Overall Officials: Partow Kebriaei, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kebriaei P, Singh H, Huls MH, Figliola MJ, Bassett R, Olivares S, Jena B, Dawson MJ, Kumaresan PR, Su S, Maiti S, Dai J, Moriarity B, Forget MA, Senyukov V, Orozco A, Liu T, McCarty J, Jackson RN, Moyes JS, Rondon G, Qazilbash M, Ciurea S, Alousi A, Nieto Y, Rezvani K, Marin D, Popat U, Hosing C, Shpall EJ, Kantarjian H, Keating M, Wierda W, Do KA, Largaespada DA, Lee DA, Hackett PB, Champlin RE, Cooper LJ. Phase I trials using Sleeping Beauty to generate CD19-specific CAR T cells. J Clin Invest. 2016 Sep 1;126(9):3363-76. doi: 10.1172/JCI86721. Epub 2016 Aug 2. PMID 27482888
- See also: MD Anderson Cancer Center — http://mdanderson.org